CLINICAL TRIAL: NCT04589000
Title: The Effect of Acupressure in Non-breastfeeding Mothers After Preterm Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Esra SARI (Other)
Responsible Party: Sponsor-Investigator, Esra SARI, Research Assistant, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: ESARI; Esra SARI (Registry Identifier: ESARI)
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Acupressure; Breastfeeding
Keywords: acupressure, breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blind. Investigator know which participant have been assigned which group but participant don't know
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure (Experimental): Throughout the study, acupressure will be applied to the acupressure group once on the post-op day 0, 2 times on the post-op 1st day, and once on the post-op 2nd day, 4 times in total for 15 minutes.
  15 minutes after acupressure application, milk will be expressed for 15 minutes and the amount of milk expressed will be recorded in the milk measurement table.
  Interventions: Other: acupressure
- control (No Intervention): No accupressure will be applied. Milk will be expressed for a total of 15 minutes, 1 time on the post-op 0th day, 2 times on the post-op 1st day and once on the post-op 2nd day for a total of 15 minutes and will be recorded in the milk measurement table.

INTERVENTIONS:
Other: acupressure — Throughout the study, acupressure will be applied to the acupressure group once on the post-op day 0, 2 times on the post-op 1st day, and once on the post-op 2nd day, 4 times in total for 15 minutes.
  15 minutes after acupressure application, milk will be expressed for 15 minutes and the amount of milk expressed will be recorded in the milk measurement table.
  Arms: acupressure

SUMMARY:
The effect of acupressure in non-breastfeeding mothers after preterm cesarean delivery

DETAILED DESCRIPTION:
One of the frequently encountered problems in breastfeeding is insufficient lactation. Numerous integrative treatments support to overcome this problem.

This randomized controlled experimental study will conduct to determine the effect of acupressure on lactation in non-breastfeeding mothers following preterm caesarean delivery.

The sample of the study will comprise of 64 mothers (32 acupressure-experimental and 32 control group), who will randomly select from among the primipara mothers of premature newborns delivered through cesarean section at Dursun Odabaş Medical Center of Van Yüzüncü Yıl University. Before the implementation, the Depression-Anxiety-Stress Scale and the Richard Campbell Sleep Quality Scale will apply. In post-operative three days, 15-minute acupressure will implement in the morning/evening, for acupressure-group mothers and pump milking will apply; control group mothers will only milked in mornings and evenings. Lactation symptoms will evaluate with Visual Analog Scale and acupressure satisfaction with Analog Patient Satisfaction Scale, and milk quantities will record.

ELIGIBILITY:
Inclusion Criteria:

* Mothers between the ages of 19-35,

  * Mothers who gave birth by cesarean operation,
  * Mothers who gave birth before 37th week of pregnancy,
  * Primiparous mothers,
  * Mothers whose baby is lying in NICU,
  * Mothers who do not have any chronic diseases,
  * Mothers who do not use breast milk enhancing drugs, vitamins and supplements,
  * Mothers who do not have any anotomic disorder in the breast,
  * Mothers who cannot breastfeed,
  * Mothers who do not have any injured skin, fracture, swelling or muscle pain, especially in the little finger.
  * Mothers without literacy problems, mental disabilities and communication problems,
  * Mothers living within the borders of the province of Van,
  * Mothers who agree to participate in the study.

Exclusion Criteria:

* Mothers of premature newborns who cannot be fed breast milk,

  * Mothers who are multiparous,
  * Mothers with chronic disease,
  * Mothers who have a condition preventing milking,
  * Mothers whose language is insufficient in understanding and speaking Turkish,
  * Mothers who have breast abscess problems,
  * Mothers who have babies with congenital anomalies,
  * They are mothers who do not volunteer to participate in the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
the amount of breast milk | 3 days
  The amount of milk will be checked twice a day 15 minutes after acupressure application

SECONDARY OUTCOMES:
The time of onset of the first colostrum and the symptoms of the first milk in mothers | 3 days
Visual Analogue Satisfaction Patient Scale (VASPS) for Breastfeeding Satisfaction | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Esra Sarı, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided